CLINICAL TRIAL: NCT03514641
Title: An Integrated Assessment of the Safety and Effectiveness of Bexagliflozin Tablets, 20 mg, for the Management of Essential Hypertension
Brief Title: An Integrated Assessment of the Safety and Effectiveness of Bexagliflozin for the Management of Essential Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-603
Record Dates: First submitted 2017-11-08; First posted 2018-05-02 (Actual); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — bexagliflozin

STUDY DESIGN:
Intervention Model Description: The primary endpoint of study 603A is the change from baseline (Day 1) to week 12 in the 24-hour average SBP of the bexagliflozin group compared to the placebo group using a superiority testing at an overall two-sided 0.05 level of significance.
  The primary endpoint of study 603B is the change from week 12 (cumulative week 24) to week 24 (cumulative week 36) in the 24-hour average SBP in the bexagliflozin group compared to the placebo group using a superiority testing at an overall two-sided 0.05 level of significance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Study 603A: bexagliflozin tablets, 20 mg or placebo
  * Study 603B week 1 to week 12: bexagliflozin tablets, 20 mg, open-labeled
  * Study 603B week 13 to week 24: bexagliflozin tablets, 20 mg or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Other): Period 1: Placebo Period 2: Bexagliflozin Period 3: Bexagliflozin
  Interventions: Drug: Bexagliflozin; Drug: Placebo
- Sequence 2 (Other): Period 1: Placebo Period 2: Bexagliflozin Period 3: Placebo
  Interventions: Drug: Bexagliflozin; Drug: Placebo
- Sequence 3 (Other): Period 1: Bexagliflozin Period 2: Bexagliflozin Period 3: Bexagliflozin
  Interventions: Drug: Bexagliflozin
- Sequence 4 (Other): Period 1: Bexagliflozin Period 2: Bexagliflozin Period 3: Placebo
  Interventions: Drug: Bexagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin tablet, 20 mg
  Other Names: EGT0001442
Drug: Placebo — Placebo (inactive) tablet to match the active drug
  Arms: Sequence 1; Sequence 2; Sequence 4

SUMMARY:
This integrated assessment consists of two studies, 603A and 603B, to be carried out sequentially in a common study population. Participating subjects informed of the trial design and their consent to participate in both studies were to be obtained in a single consent form. Approximately 680 male or female adult subjects were to be enrolled.

DETAILED DESCRIPTION:
THR-1442-C-603 is an integrated assessment of the potential utility of bexagliflozin tablets, 20 mg for the treatment of essential hypertension. It is composed of two studies, 603A and 603B, measuring effects in a common population.

603A was a multicenter double-blind parallel group placebo-controlled study conducted to determine the placebo-adjusted change from baseline to week 12 in the mean ambulatory systolic blood pressure (SBP) of approximately 680 subjects considered generally representative of the adult hypertensive population in the United States. Secondary endpoints included the placebo-adjusted change from baseline to week 12 of the mean office seated systolic blood pressure, the change to week 12 of the mean ambulatory and mean office seated diastolic blood pressure, the proportion of subjects achieving prespecified goals for absolute systolic and diastolic blood pressure as well as prespecified goals for reduction in systolic and diastolic blood pressure, measured by ambulatory and seated office measurement methodology.

A603B was a multicenter double-blind parallel group placebo-controlled randomized withdrawal study conducted to determine the durability of the antihypertensive effect of bexagliflozin tablets, 20 mg, in a population not pre-selected for existing diabetes. All subjects entered a 12 week run-in period during which they self-administered open label bexagliflozin tablets, 20 mg once daily. At week 12 a baseline ambulatory blood pressure monitoring (ABPM) measurement was made, and the subjects were randomized one to one to receive either bexagliflozin tablets, 20 mg or bexagliflozin tablets, placebo. After a 12 week treatment period a second ABPM measurement was made. The primary endpoint was the intergroup difference in the change from baseline in the mean SBP.

ELIGIBILITY:
To be eligible for randomization a prospective subject was to be:

* Male or female of age ≥ 20 years
* Diagnosed with essential hypertension and exhibiting an office seated SBP ≥ 140 and < 180 mm Hg
* Unmedicated or prescribed no more than 4 agents for hypertension. Unmedicated subjects were subjects who had never taken medications for hypertension or had not taken any anti-hypertensive medication for at least 3 months. A stable dose meant no change in dose or frequency had taken place in the 4 weeks prior to the screening visit
* If female and of childbearing potential, willing to use an adequate method of contraception and to not become pregnant for the duration of the study.
* Willing and able to return for all clinic visits and to complete all study-required procedures
* Able to self-medicate during the run-in period, omitting no more than one day of dosing
* Shown to have a seated SBP ≥ 140 and < 180 mm Hg
* Shown to exhibit a mean 24 h SBP ≥ 135 mm Hg

Prospective participants exhibiting any of the following characteristics were to be excluded from the study:

* Diagnosis of type 1 diabetes mellitus or maturity-onset/diabetes of the young (MODY)
* Known history of secondary or malignant hypertension
* Seated diastolic blood pressure (DBP) >110 mm Hg at screening
* Taking insulin for diabetes
* Prescribed more than 4 anti-hypertension medications
* Having a genitourinary tract infection within 6 weeks of screening or history of ≥ 3 genitourinary infections requiring treatment within the last 6 months
* Having cancer, active or in remission for < 3 years
* History of alcohol or illicit drug abuse in the past 2 years
* History of myocardial infarction, stroke or hospitalization for heart failure in the prior 6 months
* Previous exposure to bexagliflozin or EGT0001474
* History of hypertensive emergency
* History of sodium glucose linked transporter 2 (SGLT2) inhibitor treatment in the last 3 months
* Known intolerance or allergy to SGTL2 inhibitors
* Any condition, disease, disorder, or clinically relevant laboratory abnormality that, in the opinion of the PI, would jeopardize the subject's appropriate participation in this study or obscure the effects of treatment
* Pregnancy or nursing
* Current participation in another interventional trial or having been exposed to an investigational drug within 30 days or 7 half-lives of screening, whichever is longer
* Arm circumference too large or small to allow accurate ambulatory monitoring
* History of kidney transplant
* Occupational or other lifestyle factors that could hamper the collection of valid ABPM data
* Evidence of abnormal liver function tests (total bilirubin or alkaline phosphatase > 1.5 × upper limit of normal (ULN) with the exception of isolated Gilbert's syndrome); or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULN
* Estimated glomerular filtration rate (eGFR), as calculated by the modification of diet in renal disease study equation (MDRD), < 45 mL/min/1.73 m2 or requiring dialysis
* HbA1c > 9.5%
* Positive urine pregnancy test for female subjects of child bearing potential
* Evidence of abnormal liver function tests (total bilirubin or alkaline phosphatase > 1.5 × upper limit of normal (ULN) with the exception of isolated Gilbert's syndrome); or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULN
* eGFR, as calculated by the modification of diet in renal disease study equation (MDRD), < 45 mL/min/1.73 m2 or requiring dialysis
* HbA1c > 9.5%
* Positive urine pregnancy test for female subjects of child bearing potential

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Allegretti, M.D., Study Director — Massachusetts General Hospital
Locations (80):
- United States (80):
  - Clinical Research Site, Birmingham, Alabama
  - Clinical Research Site, Foley, Alabama
  - Clinical Research Site, Gulf Shores, Alabama
  - Clinical Research Site, Glendale, Arizona
  - Clinical Research Site, Mesa, Arizona
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Tucson, Arizona
  - Clinical Research Site, Anaheim, California
  - Clinical Research Site, Bellflower, California
  - Clinical Research Site, Fair Oaks, California
  - Clinical Research Site, Fresno, California
  - Clinical Research Site, Lincoln, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, San Gabriel, California
  - Clinical Research Site, Santa Rosa, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Colorado Springs, Colorado
  - Clinical Research Site, Denver, Colorado
  - Clinical Research Site, Golden, Colorado
  - Clinical Research Site, Stamford, Connecticut
  - Clinical Research Site, Decatur, Georgia
  - Clinical Research Site, Lithonia, Georgia
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site, Avon, Indiana
  - Clinical Research Site, Evansville, Indiana
  - Clinical Research Site, Indianapolis, Indiana
  - Clinical Research Site, Council Bluffs, Iowa
  - Clinical Research Site, Prairie Village, Kansas
  - Clinical Research Site, Lexington, Kentucky
  - Clinical Research Site, Paducah, Kentucky
  - Clinical Research Site, Versailles, Kentucky
  - Clinical Research Site, New Orleans, Louisiana
  - Clinical Research Site, Auburn, Maine
  - Clinical Research Site, Silver Spring, Maryland
  - Clinical Research Site, Edina, Minnesota
  - Clinical Research Site, Bridgeton, Missouri
  - Clinical Research Site, St Louis, Missouri
  - Clinical Research Site, Henderson, Nevada
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Trenton, New Jersey
  - Clinical Research Site, Albuquerque, New Mexico
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, Hartsdale, New York
  - Clinical Research Site, The Bronx, New York
  - Clinical Research Site, Shelby, North Carolina
  - Clinical Research Site, Akron, Ohio
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Columbus, Ohio
  - Clinical Research Site, Dayton, Ohio
  - Clinical Research Site, Dublin, Ohio
  - Clinical Research Site, Grove City, Ohio
  - Clinical Research Site, Lyndhurst, Ohio
  - Clinical Research Site, Edmond, Oklahoma
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Altoona, Pennsylvania
  - Clinical Research Site, Hatboro, Pennsylvania
  - Clinical Research Site, Lincoln, Rhode Island
  - Clinical Research Site 2, Anderson, South Carolina
  - Clinical Research Site, Anderson, South Carolina
  - Clinical Research Site, Greer, South Carolina
  - Clinical Research Site, Kingsport, Tennessee
  - Clinical Research Site, Knoxville, Tennessee
  - Clinical Research Site, Arlington, Texas
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Houston, Texas
  - Clinical Research Site, Kingwood, Texas
  - Clinical Research Site, Mesquite, Texas
  - Clinical Research Site, Plano, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Tomball, Texas
  - Clinical Research Site, Layton, Utah
  - Clinical Research Site, Murray, Utah
  - Clinical Research Site, West Jordan, Utah
  - Clinical Research Site, Arlington, Virginia
  - Clinical Research Site, Burke, Virginia
  - Clinical Research Site, Charlottesville, Virginia
  - Clinical Research Site, Danville, Virginia
  - Clinical Research Site, Manassas, Virginia
  - Clinical Research Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the first part of the study (603A), the subjects were randomized to receive bexagliflozin or placebo for 12 weeks.
Groups:
- 603A: Bexagliflozin Tablets, 20 mg: Each subject will receive bexagliflozin tablets, 20 mg once daily for 12 weeks
- 603A: Placebo Tablets: Each subject will receive placebo (inactive tablet) once daily for 12 weeks.
- 603B: Bexagliflozin Tablets, 20 mg: Each subject will receive bexagliflozin tablets, 20 mg once daily for 12 weeks from week 24 to week 36 (cumulative)
- 603B: Placebo Tablets: Each subject will receive placebo (inactive tablet) once daily for 12 weeks from week 24 to week 36 (cumulative)
Period: 603A: 0-12 Week Study Period
Arm/Group | 603A: Bexagliflozin Tablets, 20 mg | 603A: Placebo Tablets | 603B: Bexagliflozin Tablets, 20 mg | 603B: Placebo Tablets
Started | 334 | 339 | 0 | 0
Completed | 307 | 319 | 0 | 0
Not Completed | 27 | 20 | 0 | 0
Not completed — Protocol Violation | 3 | 3 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 0 | 0
Not completed — Lost to Follow-up | 10 | 9 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — 24 hr ABPM not enough readings | 0 | 1 | 0 | 0
Period: 603B: 24-36 Week Study Period
Arm/Group | 603A: Bexagliflozin Tablets, 20 mg | 603A: Placebo Tablets | 603B: Bexagliflozin Tablets, 20 mg | 603B: Placebo Tablets
Started | 0 (The second part of study only applies to subjects in 603B) | 0 (The second part of study only applies to subjects in 603B) | 281 (The subjects were re-randomized in 603B) | 281 (The subjects were re-randomized in 603B)
Completed | 0 | 0 | 267 | 266
Not Completed | 0 | 0 | 14 | 15
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 6 | 6
Not completed — 24 hr ABPM not enough readings | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: * To avoid being double-counting of the participants, the number of baseline participants has been entered as "0" for 603B.
  * Subjects in 603B study had completed 603A study and were qualified to be re-randomized in 603B study.
Groups:
- 603 A: Placebo Tablets: Each subject will receive placebo (inactive tablet) once daily for 12 weeks.
- 603B: Bexagliflozin Tablets, 20 mg: Each eligible subject who have completed 603A including two successful 24-h ABPM sessions at 603A baseline and at week 12, and have completed the 12 weeks open labeled bexagliflozin run-in period with a successful 24-h ABPM session at week 12 of 603B, will receive bexagliflozin tablets, 20 mg once daily for 12 weeks.
- 603B: Placebo Tablets: Each eligible subject who have completed 603A including two successful 24-h ABPM sessions at 603A baseline and at week 12, and have completed the 12 weeks open labeled bexagliflozin run-in period with a successful 24-h ABPM session at week 12 of 603B, will receive placebo (inactive tablets) once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | 603A: Bexagliflozin Tablets, 20 mg | 603 A: Placebo Tablets | 603B: Bexagliflozin Tablets, 20 mg | 603B: Placebo Tablets | Total
Number analyzed (Participants) | 334 | 339 | 281 | 281 | 1235
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  years
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period | 59.4 (11.32) | 58.3 (12.06) |  |  | 58.9 (11.71)
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period |  |  | 59.9 (11.39) | 59.2 (11.78) | 59.6 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  Participants
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period: Female | 127 | 139 | 0 | 0 | 266
    603A: 0-12 Week Study Period: Male | 207 | 200 | 0 | 0 | 407
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period: Female | 0 | 0 | 110 | 114 | 224
    603B: 12-36 Week Study Period: Male | 0 | 0 | 171 | 167 | 338
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  Participants
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period: Hispanic or Latino | 27 | 27 | 0 | 0 | 54
    603A: 0-12 Week Study Period: Not Hispanic or Latino | 307 | 312 | 0 | 0 | 619
    603A: 0-12 Week Study Period: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period: Hispanic or Latino | 0 | 0 | 27 | 19 | 46
    603B: 12-36 Week Study Period: Not Hispanic or Latino | 0 | 0 | 254 | 262 | 516
    603B: 12-36 Week Study Period: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  Participants
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period: American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
    603A: 0-12 Week Study Period: Asian | 7 | 4 | 0 | 0 | 11
    603A: 0-12 Week Study Period: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
    603A: 0-12 Week Study Period: Black or African American | 94 | 104 | 0 | 0 | 198
    603A: 0-12 Week Study Period: White | 219 | 220 | 0 | 0 | 439
    603A: 0-12 Week Study Period: More than one race | 4 | 3 | 0 | 0 | 7
    603A: 0-12 Week Study Period: Unknown or Not Reported | 9 | 6 | 0 | 0 | 15
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period: American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
    603B: 12-36 Week Study Period: Asian | 0 | 0 | 4 | 4 | 8
    603B: 12-36 Week Study Period: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    603B: 12-36 Week Study Period: Black or African American | 0 | 0 | 92 | 70 | 162
    603B: 12-36 Week Study Period: White | 0 | 0 | 178 | 195 | 373
    603B: 12-36 Week Study Period: More than one race | 0 | 0 | 2 | 4 | 6
    603B: 12-36 Week Study Period: Unknown or Not Reported | 0 | 0 | 4 | 7 | 11
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  kg/m^2
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period | 32.29 (6.522) | 32.90 (6.527) |  |  | 32.59 (6.527)
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period |  |  | 32.22 (6.952) | 33.17 (6.144) | 32.69 (6.572)
Body Weight at Baseline [Mean (Standard Deviation); unit: kg] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  kg
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period | 95.36 (22.643) | 97.47 (22.673) |  |  | 96.42 (22.666)
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period |  |  | 95.71 (24.321) | 97.55 (21.003) | 96.63 (22.721)
History of Diabetes [Count of Participants; unit: Participants] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  Participants
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period: Yes | 83 | 84 |  |  | 167
    603A: 0-12 Week Study Period: No | 251 | 255 |  |  | 506
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period: Yes |  |  | 78 | 66 | 144
    603B: 12-36 Week Study Period: No |  |  | 203 | 215 | 418
Use of any antihypertension medication [Count of Participants; unit: Participants] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  Participants
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period | 269 | 276 |  |  | 545
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period |  |  | 233 | 226 | 459
Estimated Glomerular Filtration Rate (eGFR) Mean [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  mL/min/1.73 m^2
    603A: 0-12 Week Study Period: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period | 82.64 (17.438) | 84.42 (19.710) |  |  | 83.53 (18.625)
    603B: 12-36 Week Study Period: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period |  |  | 78.75 (18.971) | 77.95 (18.871) | 78.35 (18.908)
Ambulatory Blood Pressure Monitoring (ABPM) at baseline [Mean (Standard Deviation); unit: mm Hg] — Population: Subjects who experienced worsening of their hypertension prior to the 6-week visit were not to undergo ABPM measurement.
  mm Hg
    603A: 0-12 Week Study Period; SBP: number analyzed (Participants) | 329 | 339 | 0 | 0 | 668
    603A: 0-12 Week Study Period; SBP | 147.58 (9.640) | 147.48 (10.064) |  |  | 147.53 (9.850)
    603A: 0-12 Week Study Period; DBP: number analyzed (Participants) | 329 | 339 | 0 | 0 | 668
    603A: 0-12 Week Study Period; DBP | 85.04 (9.240) | 84.97 (10.216) |  |  | 85.01 (9.740)
    603B: 12-36 Week Study Period; SBP: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period; SBP |  |  | 136.30 (13.844) | 135.62 (13.510) | 135.96 (13.67)
    603B: 12-36 Week Study Period; DBP: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period; DBP |  |  | 79.58 (10.471) | 79.20 (10.571) | 79.39 (10.513)
Office seated SBP and DBP at baseline [Mean (Standard Deviation); unit: mm Hg] — Population: First row corresponds to participants only in 603A. Second row corresponds to participants only in 603B.
  mm Hg
    603A: 0-12 Week Study Period; SBP: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period; SBP | 156.44 (10.513) | 155.84 (10.335) |  |  | 156.14 (10.420)
    603A: 0-12 Week Study Period; DBP: number analyzed (Participants) | 334 | 339 | 0 | 0 | 673
    603A: 0-12 Week Study Period; DBP | 91.29 (10.269) | 91.48 (10.619) |  |  | 91.39 (10.439)
    603B: 12-36 Week Study Period; SBP: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period; SBP |  |  | 141.18 (16.231) | 140.69 (14.960) | 140.94 (15.596)
    603B: 12-36 Week Study Period; DBP: number analyzed (Participants) | 0 | 0 | 281 | 281 | 562
    603B: 12-36 Week Study Period; DBP |  |  | 84.75 (11.623) | 85.28 (11.588) | 84.55 (10.985)

OUTCOME MEASURES:

1. Primary Outcome: Change of the 24 Hour Mean Systolic Blood Pressure From Baseline (Day 1) to Week 12
Description: Change of the 24 hour mean systolic blood pressure in the bexagliflozin group compared to placebo
Time Frame: Baseline (Day 1) to week 12
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Bexagliflozin Tablets, 20 mg: Each subject will receive bexagliflozin tablets, 20 mg once daily for 12 weeks.
- Placebo Tablets: Each subject will receive placebo (inactive tablet) once daily for 12 weeks.
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
mm Hg | -8.86 (0.642) | -6.15 (0.622)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0025, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; LS Means difference = -2.72, 95% CI 2-sided [-4.47 to -0.96]

2. Primary Outcome: Change of the 24 Hour Mean Systolic Blood Pressure From Cumulative Week 24 to Week 36
Description: Change of the 24 hour mean systolic blood pressure in the bexagliflozin group compared placebo
Time Frame: Change from week 24 to week 36
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 281 | 281
mm Hg | 0.30 (0.680) | 2.74 (0.678)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0117, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-4.32 to -0.54]

3. Secondary Outcome: 603A, Reduction of Mean Ambulatory Systolic Blood Pressure
Description: Proportion of subjects who achieve a reduction of mean ambulatory systolic blood pressure of 10 mm Hg or greater
Time Frame: Baseline (Day 1) to week 12
Population: The full model is a logistic regression that includes diabetes status (history of type 2 diabetes mellitus or not), eGFR at screening, pre-treatment status (presently medicated for hypertension or not), treatment, and the baseline 24-hour mean SBP/DBP value as a fixed effect covariate.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
proportion of participants | 0.40 [0.35 to 0.46] | 0.34 [0.29 to 0.40]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.1317, Covariance — Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.92 to 1.83]

4. Secondary Outcome: 603A, Mean Ambulatory Systolic Blood Pressure of 135 mm Hg or Less
Description: Proportion of subjects who achieve a mean ambulatory systolic blood pressure of 135 mm Hg or less
Time Frame: Baseline (Day 1) to week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
Proportion of subjects | 0.40 [0.34 to 0.46] | 0.29 [0.24 to 0.35]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0113, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.11 to 2.30]

5. Secondary Outcome: 603A, Change in Seated Office Systolic Blood Pressure
Description: Placebo-adjusted change in seated office systolic blood pressure
Time Frame: Baseline (Day 1) to week 12
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
mm Hg | -11.24 (0.799) | -6.61 (0.787)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p < 0.0001, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Mean Difference (Final Values) = -4.63, 95% CI 2-sided [-6.83 to -2.42]

6. Secondary Outcome: 603A, Seated Office Systolic Blood Pressure of 140 mm Hg or Less
Description: Proportion of subjects who achieve a seated office systolic blood pressure of 140 mm Hg or less
Time Frame: Baseline (Day 1) to week 12
Population: The full model is a logistic regression that includes diabetes status (history of type 2 diabetes mellitus or not), eGFR at screening, pre-treatment status (presently medicated for hypertension or not), treatment, and the baseline seated office SBP/DBP value as a fixed effect covariate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
Proportion of subjects | 0.38 [0.33 to 0.44] | 0.25 [0.21 to 0.30]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0004, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.32 to 2.62]

7. Secondary Outcome: 603A, Change in Mean Ambulatory Diastolic Blood Pressure
Description: Placebo-adjusted change in mean ambulatory diastolic blood pressure
Time Frame: Baseline (Day 1) to week 12
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
mm Hg | -3.92 (0.349) | -3.08 (0.337)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0863, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.79 to 0.12]

8. Secondary Outcome: 603A, Mean Ambulatory Diastolic Blood Pressure of 87 mm Hg or Less
Description: Proportion of subjects who achieve a mean ambulatory diastolic blood pressure of 87 mm Hg or less
Time Frame: Baseline (Day 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
Proportion of subjects | 0.47 [0.41 to 0.53] | 0.37 [0.32 to 0.43]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0232, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.06 to 2.08]

9. Secondary Outcome: 603A, Reduction of Mean Ambulatory Diastolic Blood Pressure of 4 mm Hg or Greater
Description: Proportion of subjects who achieve a reduction of mean ambulatory diastolic blood pressure of 4 mm Hg or greater
Time Frame: Baseline (Day 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
Proportion of subjects | 0.88 [0.83 to 0.92] | 0.80 [0.73 to 0.85]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0140, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.13 to 2.91]

10. Secondary Outcome: 603A, Change in Seated Office Diastolic Blood Pressure
Description: Placebo-adjusted change in seated office diastolic blood pressure
Time Frame: Baseline (Day 1) to week 12
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
mm Hg | -4.44 (0.504) | -2.13 (0.496)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0011, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Mean Difference (Final Values) = -2.31, 95% CI 2-sided [-3.70 to -0.92]

11. Secondary Outcome: 603A, Seated Office Diastolic Blood Pressure of 90 mm Hg or Less
Description: Proportion of subjects who achieve a mean seated office diastolic blood pressure of 90 mm Hg or less
Time Frame: Baseline (Day 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 334 | 339
Proportion of subjects | 0.65 [0.59 to 0.71] | 0.53 [0.47 to 0.59]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0094, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.13 to 2.35]

12. Secondary Outcome: 603B, Change in Seated Office Systolic Blood Pressure
Description: Placebo-adjusted change from week 12 to week 24 in seated office systolic blood pressure
Time Frame: Week 12 (cumulative week 24) to Week 24 (cumulative week 36)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 281 | 281
mm Hg | 1.98 (0.846) | 5.18 (0.859)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0083, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-5.57 to -0.83]

13. Secondary Outcome: 603B, Change in Mean Ambulatory Diastolic Blood Pressure
Description: Placebo-adjusted change in mean ambulatory diastolic blood pressure
Time Frame: Week 12 (cumulative week 24) to Week 24 (cumulative week 36)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 281 | 281
mm Hg | 0.10 (0.369) | 0.94 (0.368)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.1085, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.87 to 0.19]

14. Secondary Outcome: 603B, Change in Seated Office Diastolic Blood Pressure
Description: Placebo-adjusted change from week 12 to week 24 in seated office diastolic blood pressure
Time Frame: Week 12 (cumulative week 24) to Week 24 (cumulative week 36)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 281 | 281
mm Hg | 0.51 (0.507) | 1.76 (0.514)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0837, Covariance; Covariance model diabetes status, eGFR at screening, pre-treatment status, treatment, and baseline 24-hour mean SBP; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-2.67 to 0.17]

15. Other Pre Specified Outcome: Integrated 603A and 603B, Effects on Mean Ambulatory Systolic and Diastolic Blood Pressure
Description: Integration of measures collected in studies 603A and 603B will be used to assess consistent effects on mean ambulatory systolic and diastolic blood pressure after 12 weeks of bexagliflozin treatment, as well as longer treatment periods, i.e., 24 weeks or 36 weeks of bexagliflozin treatment.
Time Frame: Baseline (Day 1) to cumulative week 36
Population: Number of subjects with baseline and value after specified weeks of exposure to Bexagliflozin
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Effect on Mean Ambulatory SBP: Effect on ABPM SBP after 12, 24, and 36 weeks of cumulative exposure to Bexagliflozin
- Effect on Mean Ambulatory DBP: Effect on ABPM DBP after 12, 24, and 36 weeks of cumulative exposure to Bexagliflozin
Arm/Group | Effect on Mean Ambulatory SBP | Effect on Mean Ambulatory DBP
Number analyzed (Participants) | 649 | 649
mm Hg
  12 Weeks: number analyzed (Participants) | 649 | 555
  12 Weeks | -7.595 [-8.565 to -6.625] | -3.269 [-3.773 to -2.764]
  24 Weeks: number analyzed (Participants) | 395 | 395
  24 Weeks | -9.262 [-10.559 to -7.965] | -4.044 [-4.720 to -3.368]
  36 Weeks: number analyzed (Participants) | 119 | 119
  36 Weeks | -12.454 [-14.988 to -9.921] | -5.566 [-6.825 to -4.308]

16. Other Pre Specified Outcome: Integrated 603A and 603B, Effects on Seated Office Systolic and Diastolic Blood Pressure
Description: Integration of measures collected in studies 603A and 603B will be used to assess consistent effects on seated office systolic and diastolic blood pressure over time
Time Frame: Baseline (Day 1) to cumulative week 36
Population: Number of subjects with baseline and value after specified weeks of exposure to Bexagliflozin
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Effect on Seated Office SBP: Effect on seated office SBP after 6, 12, 18, 24, and 36 weeks of cumulative exposure to Bexagliflozin
- Effect on Seated Office DBP: Effect on seated office DBP after 6, 12, 18, 24, and 36 weeks of cumulative exposure to Bexagliflozin
Arm/Group | Effect on Seated Office SBP | Effect on Seated Office DBP
Number analyzed (Participants) | 649 | 649
mm Hg
  6 Weeks: number analyzed (Participants) | 602 | 602
  6 Weeks | -8.43 (16.399) | -4.50 (9.534)
  12 Weeks: number analyzed (Participants) | 582 | 582
  12 Weeks | -9.91 (15.777) | -4.10 (9.716)
  18 Weeks: number analyzed (Participants) | 273 | 273
  18 Weeks | -14.46 (16.000) | -5.87 (9.282)
  24 Weeks: number analyzed (Participants) | 411 | 411
  24 Weeks | -12.53 (18.830) | -4.92 (10.910)
  36 Weeks: number analyzed (Participants) | 127 | 127
  36 Weeks | -15.71 (16.975) | -6.47 (9.933)

ADVERSE EVENTS:
Time Frame: For 603A, adverse events were collected from baseline to Week 12. For 603B, adverse events were collected from Week 24 to Week 36.
Groups:
- 603B: Placebo Tablets: Each eligible subject who have completed 603A including two successful 24-h ABPM sessions at 603A baseline and at week 12, and have completed the 12 weeks open labeled bexagliflozin run-in period with a successful 24-h ABPM session at week 12 of 603B, will receive placebo tablets (inactive), 20 mg once daily for 12 weeks.
Arm/Group | 603A: Bexagliflozin Tablets, 20 mg | 603A: Placebo Tablets | 603B: Bexagliflozin Tablets, 20 mg | 603B: Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 0/334 | 0/339 | 0/281 | 0/281
Serious Adverse Events (participants affected / at risk) | 11/334 | 10/339 | 9/281 | 6/281
Other Adverse Events (participants affected / at risk) | 94/334 | 88/339 | 32/281 | 37/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 603A: Bexagliflozin Tablets, 20 mg (N=334) | 603A: Placebo Tablets (N=339) | 603B: Bexagliflozin Tablets, 20 mg (N=281) | 603B: Placebo Tablets (N=281)
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle rupture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 603A: Bexagliflozin Tablets, 20 mg (N=334) | 603A: Placebo Tablets (N=339) | 603B: Bexagliflozin Tablets, 20 mg (N=281) | 603B: Placebo Tablets (N=281)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (7) | 3 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 7 (7) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Genital infection fungal (Infections and infestations) | 4 (8) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (12) | 11 (11) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 10 (11) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 7 (7) | 7 (7) | 6 (6) | 6 (7)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 1 (1) | 2 (2)
Polydipsia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 1 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 7 (7) | 1 (1) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 7 (7) | 1 (1) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 13 (13) | 4 (4) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 4 (4) | 9 (9) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 6 (6) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator has no right to publish the study results.

DOCUMENTS (2):
  • Study Protocol (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03514641/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT03514641/SAP_001.pdf